CLINICAL TRIAL: NCT00042055
Title: A Phase II Pilot Study of CP-461 in the Treatment of Moderately to Severely Active Crohn's Disease
Brief Title: CP-461 for the Treatment of Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Cell Pathways (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-461-012
Record Dates: First submitted 2002-07-22; First posted 2002-07-24 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — (5-fluoro-2-methyl-1-(4-pyridyl)methylene-3-(N-benzyl)-indene)-acetamide hydrochloride

INTERVENTIONS:
Drug: CP-461

SUMMARY:
Patients with moderately to severely active Crohn's disease will be treated with oral CP-461 200 mg (2 x 100 mg capsules) twice-daily for 8 weeks.

The purpose of this study is to see if CP-461 improves the symptoms of Crohn's disease and/or the patient's quality of life. Patient's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > or = 18 years of age.
* Crohn's Disease Activity Index (CDAI) of > or = 220 and < or = 400.
* Crohn's disease of at least 3 months duration with colitis, ileitis, or ileocolitis, confirmed by radiography or endoscopy.
* Men and women of childbearing potential must use adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization).
* Concomitant medications:

  * If using aminosalicylates, the patient must have been using the aminosalicylates for at least 2 months before pre-screening. The dose must be stable for at least 2 weeks before pre-screening. If aminosalicylates are to be discontinued, it must be done at least 2 weeks before pre-screening.
  * If using oral corticosteroids, the patient must have been receiving them for at least 2 months and must be on a stable dosage (< or = 40 mg/day prednisone equivalent) for at least 2 weeks before pre-screening.
  * If using infliximab, the patient must not have received an infliximab infusion for at least 12 weeks.
  * If using azathioprine, 6-mercaptopurine (6-MP), or mycophenolate mofetil, the start date must be at least 3 months prior to pre-screening and the dose must be stable for at least 8 weeks before pre-screening.
  * If using methotrexate, the patient must have been using methotrexate for at least 4 months before pre-screening with a stable dosage of at least 6 weeks.
  * If using Crohn's disease-specific antibiotics, the patient must have been using them for at least 2 weeks at a stable dosage.
* The screening laboratory tests must meet the following criteria:

  * Hemoglobin > or = 8.5
  * WBC > or = 3.5 x 10 9/L
  * Neutrophils > or = 1.5 x 10 9/L
  * Platelets > or = 100 x 10 9/L
  * Serum creatinine less than 2.2 mg/dL.
  * Transaminases (AST/ALT) must be < or = 1.5 times the upper limit of normal range for the laboratory conducting the test.
  * Bilirubin must be WNL.
* Patient must be able to adhere to the study visit schedule and other protocol requirements.
* The patient must be capable of giving informed consent and the consent must be obtained before any study specific screening procedures.

Exclusion Criteria:

* Local manifestations of Crohn's disease such as strictures, abscesses, or other disease complications for which surgery might be indicated. Conditions that might preclude utilization of CDAI to assess response to therapy (such as "short gut" syndrome). If abscess is present, it should be drained before pre-screening, with at least 3 weeks between drainage of the abscess and pre-screening.
* Positive stool culture for enteric pathogens, pathogenic ova or parasites or Clostridium difficile toxin.
* Pregnancy, nursing, or unwillingness to comply with birth control.
* Patients who are currently receiving or have been treated with cyclosporine, tacrolimus, or sirolimus within 4 weeks of pre-screening.
* Infliximab infusion within 12 weeks of pre-screening.
* Rectally administered steroids within 2 weeks of pre-screening.
* Treatment with parenteral nutrition (TPN) within 3 weeks of prescreening.
* Signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* Presence of a transplanted organ.
* Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* Known substance abuse (drug or alcohol) during the last two years.
* Patients with a fever > or = 100.5 degrees F.
* The patient is unable to return for follow-up evaluation.
* The patient has received an investigational drug or device within 30 days before the initiation of therapy.
* Refusal to sign the informed consent.
* The patient is, in the opinions of the investigators, not an appropriate candidate for the study.
* The following laboratory abnormalities:

  * Hemoglobin < 8.5
  * WBC < 3.5 x 10 9/L
  * Neutrophils < 1.5 x 10 9/L
  * Platelets < 100 x 10 9/L
  * Serum creatinine > or = 2.2 mg/dL
  * Transaminases (AST/ALT) > 1.5 times the upper limit of normal range for the laboratory conducting the test.
  * Bilirubin > upper limit of normal range for the laboratory conducting the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-07; Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Southern Drug Research, Birmingham, Alabama
  - Community Clinical Trials, Orange, California
  - Florida Medical Research Institute, PA, Gainesville, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indianapolis Gastroenterology and Hepatology, Inc., Indianapolis, Indiana
  - Digestive Disease Associates, PA, Columbia, Maryland
  - Atlantic Gastroenterology Associates, Egg Harbor, New Jersey
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Consultants for Clinical Research, Inc., Cincinnati, Ohio